CLINICAL TRIAL: NCT00364468
Title: A Randomized Dose Finding Study of KRN125 (Pegfilgrastim) for the Treatment of Chemotherapy - Induced Neutropenia in Malignant Lymphoma
Brief Title: Dose Finding Study of KRN125 (Pegfilgrastim) for Treatment of Neutropenic Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kyowa Kirin Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KRN125/05-A04
Record Dates: First submitted 2006-08-14; First posted 2006-08-15 (Estimated); Last update posted 2017-03-03 (Actual); Status verified 2017-02

CONDITIONS: Neutropenia
Keywords: pegfilgrastim; neutropenia; cancer patients; lymphoma
MeSH Terms: conditions — Neutropenia; Lymphoma | interventions — pegfilgrastim

INTERVENTIONS:
Drug: pegfilgrastim

SUMMARY:
To assess the duration of severe neutropenia in cycle 1 of chemotherapy after treatment with a single injection of KRN125 or multiple daily injections of filgrastim.

ELIGIBILITY:
Inclusion Criteria:

* patients diagnosed as malignant lymphoma
* patients who were refractory to anthracycline or anthraquinone containing chemotherapy
* patients who are going to receive ESHAP or CHASE treatment regimen
* ECOG performance status =< 2
* patients who have appropriate bone marrow, hepatic and renal functions
* written informed consent

Exclusion Criteria:

* double cancer
* history of bone marrow transplantation or PBSCT
* more than 2 prior chemotherapy regimens
* primary hematologic disease such as myelodysplastic syndrome
* previous radiotherapy within 4 weeks of enrollment
* woman of childbearing potential who were either pregnant, breast feeding
* patients who participated in other clinical trials within the last 4 weeks of enrollment

Ages: 20 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2006-03; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
To compare the duration of severe neutropenia

CONTACTS AND LOCATIONS:
Overall Officials: Tomomitsu Hotta, MD, Study Chair — Nagoya Medical Center
Locations (6):
- Japan (6):
  - Tokai region, Aichi
  - Kyusyu region, Fukuoka, Nagasaki
  - Kanto region, Gunma, Saitama, Tokyo, Kanagawa
  - Hokkaido region, Hokkaido
  - Kinki region, Kyoto, Mie, Shiga
  - Tohoku region, Miyagi